CLINICAL TRIAL: NCT06003725
Title: The Cultural Adaptation of an Alcohol and Other Drug Use Treatment for Black Justice Involved Youth
Brief Title: Cultural Adaptation of Drug Treatment for DJJ Youth
Acronym: CAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-40126; K23DA057412 (NIH)
Record Dates: First submitted 2023-07-18; First posted 2023-08-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Substance Use
Keywords: Substance use; substance misuse; adolescent; cultural adaptation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Individual interviews with Black justice-involved youth (JIY) and focus groups with guardians of Black JIY and community members will be conducted. Data from focus groups and interviews will be used to inform the cultural adaptation of an evidence-based adolescent substance use treatment. The cultural adapted treatment will then be piloted with 30 Black JIY for feasibility and acceptability.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADAP-ITT Phase 8 (Experimental): Phase 8 consists of piloting the culturally adapted CYT intervention with 30 Black JIY to examine feasibility and acceptability.
  Interventions: Behavioral: Culturally Adapted Adolescent Substance Use Treatment

INTERVENTIONS:
Behavioral: Culturally Adapted Adolescent Substance Use Treatment — The Cannabis Youth Treatment Series (CYT) (MET/CBT12 model) aims to reduce alcohol and cannabis use.
  Other Names: Cannabis Youth Treatment Series

SUMMARY:
This project aims to improve the understanding of the impact of Ethnic and Racial Discrimination (ERD) on adolescent alcohol and other drug use (AOD) within the Black Justice-Involved Youth (JIY) population. Individual interviews with Black JIY and focus groups with parents and guardians of Black JIY and community members who support change and reform in the justice community for Black JIY will be conducted.

DETAILED DESCRIPTION:
Black JIY are overrepresented in the criminal justice system due to institutional racism and discrimination. The General Strain Theory posits that high levels of ethnic and racial discrimination (ERD), paired with elevated levels of witnessing or experiencing police brutality, places Black JIY at unique risk of increased alcohol and other drug use (AOD) as a means of coping with stressful events. Black JIY report engaging in comorbid alcohol and cannabis use to achieve temporary respite from discrimination-induced stress. While JIY engage in higher rates of comorbid alcohol and cannabis use compared to non-justice-involved youth, overall, Black JIY are less likely to be diverted to substance use treatment programs, less likely to engage in care after being released on probation, less likely to benefit from substance use treatment in terms of reduced risk of recidivism, and are more adversely affected by early onset of AOD activity than White JIY. To date, no known adolescent substance use treatment directly addresses ERD, the increased risk of AOD due to ERD, or explicitly presents tools on how to appropriately respond to AOD and discrimination distress among Black JIY. To address this problem, the investigator's research program aspires to improve the understanding of the impact of ERD on adolescent AOD within the Black JIY population. Individual interviews with Black JIY and focus groups with guardians of Black JIY and community members will be conducted. Data will be used to culturally adapt an adolescent substance use intervention. The culturally adapted intervention will then be piloted with 30 Black JIY.

ELIGIBILITY:
For Focus Groups and Interviews:

Black JIY Participants:

Inclusion Criteria:

• 1) Between the ages of 13-17; 2) identify as Black or African American; and 3) on community probation.

Exclusion Criteria:

• Will be excluded if they do not have parental consent to participate.

For Focus Groups and Interviews:

Adult Participants

Inclusion Criteria:

* A guardian of JIY
* An advocate (someone who supports change and reform in the justice community) for Black JIY.

Exclusion Criteria:

• Will be excluded if they do not provide consent to participate.

For pilot feasibility study:

Black JIY Participants:

Inclusion Criteria:

* Between the ages of 13 and 17
* Identify as Black or African American
* Be on community probation
* Meet criteria for alcohol, cannabis, or other drug misuse as defined by the DSM 5
* Be experiencing at least 1 problem related to AOD;
* The frequency of AOD must be weekly use over a 3-month period

Exclusion Criteria:

* Will be excluded if they do not have parental consent to participate
* Parole violation

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability | After study completion, an average of 3 months
  Participants will complete feasibility and acceptability questionnaires and provide qualitative data on likes and dislikes about the intervention, delivery, session structure, and content.

SECONDARY OUTCOMES:
Change in substance use | Baseline, after each study visit, at study completion, up to 3 months post-intervention, an average of 6 months.
  Participants will complete urinalysis
Change in mental health symptoms | Baseline, after each study visit, at study completion, up to 3 months post-intervention, an average of 6 months.
  Participants will complete measures and questionnaires to monitor anxiety, depression, and trauma symptoms
Change in discrimination distress | baseline, after study completion, and up to 3 months post-intervention, an average of 6 months.
  Participants will complete a discrimination distress assessment measure

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Bryant, DSW, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No